CLINICAL TRIAL: NCT01836107
Title: Cross-cultural Adaptation and Validation of a Score for Evaluating Quality of Inpatient Clinical Notes
Brief Title: Adaptation and Validation of a Score From English to Spanish for Evaluating Quality of Clinical Notes
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Diego Hernan Giunta, MD, Coordinator, Hospital Italiano de Buenos Aires
Other Study IDs: 2027
Record Dates: First submitted 2013-04-08; First posted 2013-04-19 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2013-04

CONDITIONS: Validation Studies; Cross-Cultural Comparison; Medical Records; Total Quality Management
Keywords: Clinical notes; Communication between physicians; Quality; Cross-cultural adaptation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to make a Spanish version of a score that evaluates the characteristics of a good quality clinical note for the purpose of physician communication. The score is an instrument, originally made in English. Due to the score will be used in a different country, language and culture of the original protocol, it is necessary apply a process of translation and adaptation to the context where the score is going to be applied.

The process of validation implies to evaluate if the instrument produces the same results under similar conditions and if the instrument maintains the ability to measure the same features or characteristics according to the original design.

DETAILED DESCRIPTION:
Communication between health care providers is an important factor for the continuity of patient care. In the medical records, narrative components, such as clinical notes become important for this purpose. The inappropriate use of features , such as copy & paste, produces "unreadable" documents, with redundant information, reducing the quality of them. Within this framework, it is essential to assess the quality of clinical notes to implement mechanisms to improve it.

This study proposes to make a Spanish version of the Physician Documentation Quality Instrument (PDQI9) The original instrument evaluates the characteristics of a good quality clinical note for the purpose of physician communication. Due to a measuring instrument should be reliable and valid, not only for the original research population, and the score will be used in a different country, language and culture it is necessary a cross-cultural validation of the score.

The objective is to do a cross-cultural adaptation and validation of the Spanish version of "PDQI9" score, analyzing the use of PDQI-9 in a different language (Spanish), in an institution of different size (Hospital Italiano de Buenos Aires), with a different Electronic Health Record (EHR).

The process of cross-cultural validation involves two phases: the first phase is the translation and cross-cultural adaptation of the instrument. This phase will produce a Spanish version of the score and involves an expert panel of internal medicine physicians and a group of internal medicine physicians for the pilot evaluation.

The second phase evaluates the reliability and validity of the Spanish version. This phase includes internal consistency, intra-rater reliability, inter-rater reliability and the evaluation of the criterion validity of the adapted instrument. The validity of the adapted instrument will be measured comparing the score results with the Gold Standard represented by an expert committee. For every phase, the clinical notes (admission notes, progress notes and discharge summaries) will be randomly and stratified selected.

ELIGIBILITY:
Inclusion Criteria:

* For every phase, the clinical notes will be randomly and stratified selected. The clinical notes must belong to patients hospitalized at Internal Medicine area in Hospital Italiano de Buenos Aires (HIBA) without any referral to or from other medical areas. The length of stay expected should be at least three days, and the Electronic Health Record (EHR) has to contain the admission notes, progress notes and discharge summaries.

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinical notes (admission notes, progress notes and discharge summaries) will be included in the study following the original research.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Cross cultural validity of a score | 3 months
  Evaluation of criterion validity (Gold Standard vs the use of the adapted score)

CONTACTS AND LOCATIONS:
Overall Officials: Sonia E Benitez, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Buenos Aires, Argentina